CLINICAL TRIAL: NCT00796887
Title: Phase II, Randomized, Double-Blinded, Placebo-Controlled Trial of Extended-Release Niacin (Niaspan®) to Augment Subacute Ischemic Stroke Recovery
Brief Title: Randomized, Controlled Trial of Extended-Release Niacin (Niaspan®) to Augment Subacute Ischemic Stroke Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Andrew N. Russman, Senior Staff Neurologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HFHS-5284
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Recovery of Function; Extended-release niacin
MeSH Terms: conditions — Ischemic Stroke | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Niaspan® 500mg (Experimental)
  Interventions: Drug: Extended-Release Niacin
- Niaspan® 1000mg (Experimental)
  Interventions: Drug: Extended-Release Niacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended-Release Niacin — 500mg tablet once daily
  Other Names: Niaspan®
  Arms: Niaspan® 500mg
Drug: Extended-Release Niacin — 1000mg tablet once daily
  Other Names: Niaspan®
  Arms: Niaspan® 1000mg
Drug: Placebo — Placebo tablet once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and to explore the possible benefit of extended-release niacin (Niaspan®) in attempting to improve the recovery of patients after ischemic stroke.

DETAILED DESCRIPTION:
The investigators are interested in extended-release niacin (Niaspan®) and its potential restorative role after ischemic stroke. At Henry Ford Hospital in Detroit, Michigan, extended-release niacin (Niaspan®) has been shown to improve the functional outcomes of rats when administered during the first two weeks after ischemic stroke onset. Such results are encouraging and warrant further investigation in humans. The specific aims of this study are to prospectively evaluate the use of extended-release niacin (Niaspan®) in a phase II clinical trial in patients with subacute ischemic stroke. The investigators will assess the safety and tolerability of Niaspan® and evaluate outcomes among treated patients at 24 weeks after ischemic stroke onset. This will be a randomized, double-blinded, placebo-controlled, safety, tolerability, and exploratory efficacy study of extended-release niacin (Niaspan®) in subacute ischemic stroke patients with both low HDL-C and normal HDL-C in cohort sizes of 16 patients. A total enrollment of 48 patients is planned. Patients who are between 72 hours and 7 days from stroke onset will receive Niaspan® 500mg, 1000mg, or placebo daily for a period of 24 weeks. Evaluation of potential safety and tolerability in subacute ischemic stroke patients will be made during the course of treatment and at formal visits at 6, 12, and 24 weeks. The primary safety measures will be death, recurrent stroke, myocardial infarction, and neurological worsening during treatment. Exploratory analysis will include functional outcomes on the NIHSS scores, modified Rankin scores, and Barthel indices at 24 weeks. The goal of this study is to improve the outcomes from ischemic stroke, using a safe and effective novel strategy of restoration, which has been translated from basic laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical ischemic stroke able to enroll between 72 hours and 7 days after symptom onset.
* Patients age 18-85, inclusive.
* NIHSS score of 4-21, inclusive, prior to treatment.
* Signed IRB-approved informed consent by patient or authorized representative.

Exclusion Criteria:

General

* Participation in another study with an investigational drug or device.
* Women known to be pregnant, lactating, or of childbearing potential with a positive urine beta-HCG.
* Patients using niacin within the 7 days previous to their stroke.

Safety Related

* Unstable angina.
* Acute Myocardial infarction.
* Concurrent arterial bleeding.
* Active peptic ulcer disease.
* Platelet count less than 100,000 per microliter.
* Internationally Normalized Ratio (INR) greater than 1.3 without use of warfarin.
* Concurrent use of bile acid sequestrants (colestipol and cholestyramine)
* Baseline systolic blood pressure less than 100 mmHg.
* History of significant hepatic dysfunction.
* Allergy or hypersensitivity to aspirin.
* Concurrent use of amiodarone, gemfibrozil, fibrate or other bile acid resin, cyclosporine, itraconazole, ketaconazole, telithromycin, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, danazol.
* Allergy or hypersensitivity to extended-release niacin.
* Allergy or hypersensitivity to statin agents.

Potentially Interfering with Outcomes Assessment

* Prior history of dementia.
* Patients without fixed address or those deemed unlikely to present for follow-up by the investigator.
* Patients whose life expectancy is less than 24 weeks.
* Pre-stroke modified Rankin score>2.
* Glucose less than 50 mg/dl.
* Other serious illness (e.g., severe hepatic, cardiac, or renal failure; or a complex disease that may confound treatment assessment).

Imaging Related

* Evidence of primary intra-parenchymal hemorrhage on initial neuroimaging study.
* Neuroimaging evidence of a nonvascular cause for the neurological symptoms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of expected serious adverse events | 24 weeks
  Analysis of the frequency and type of serious adverse events among patients in each study arm

SECONDARY OUTCOMES:
Functional Recovery | 24 weeks
  Exploratory efficacy analysis of the differences in functional recovery between each study arm as measured using the modified Rankin Scale, NIH Stroke Scale, and Barthel Index.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N. Russman, D.O., Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States